CLINICAL TRIAL: NCT02940470
Title: Weight Loss Pilot Study in Postmenopausal Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UMN999; U54CA116849 (NIH); CPRC#2008NTLS107 (Other: University of Minnesota Cancer Protocol Review Committee)
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer; Obesity; Overweight
MeSH Terms: conditions — Breast Neoplasms; Obesity; Overweight | interventions — Caloric Restriction; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calorie restricted diet plus exercise (Experimental): See Intervention Description
  Interventions: Other: Calorie restricted diet plus exercise
- Weight management classes (Active Comparator): See Intervention Description
  Interventions: Other: Weight management classes

INTERVENTIONS:
Other: Calorie restricted diet plus exercise — Daily meals plus exercise providing 1000 kcal restriction per day for 12 weeks.
  Arms: Calorie restricted diet plus exercise
Other: Weight management classes — Weekly 1-hour weight management classes for 12 weeks.
  Arms: Weight management classes

SUMMARY:
The primary objective of this pilot study is to determine the effect of weight loss on a wide range of biomarkers associated with risk of breast cancer recurrence in overweight and obese breast cancer survivors. We hypothesized that weight loss would result in a statistically significant improvement in biomarkers associated with risk of breast cancer recurrence.

DETAILED DESCRIPTION:
Women who are overweight, obese or gain weight after a breast cancer diagnosis are at greater risk for recurrence and death compared with lighter women. There have been a few studies examining the effects of different interventions on weight loss in breast cancer survivors but very few have examined the effect of weight loss interventions on circulating levels of markers associated with cancer risk. The overall objective of this proposal is to determine how weight loss affects circulating levels of biomarkers associated with breast cancer risk and recurrence, and quality of life of overweight and obese breast cancer survivors. The central hypothesis is that weight loss will decrease the levels of markers adversely associated with breast cancer and increase quality of life in these women. To test the central hypothesis the following specific aims will be pursued:

* To assess the effects of two different weight loss interventions on biomarkers associated with breast cancer risk and recurrence
* To assess the impact of the weight loss interventions on quality of life and sleep
* To assess the impact of weight loss on measures of bone health

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal (defined as experiencing at least 12 months without a menstrual period)
* diagnosed with operable invasive breast cancer and treated with mastectomy or with lumpectomy and radiation
* completed all surgery, radiation, and systemic chemotherapy one to 12 months prior to enrollment
* BMI ≥ 27 kg/m2
* less than 7 servings of alcohol per week
* willing to be randomized into either group
* not planning to move away from the area during the period of study
* non-smoker

Exclusion Criteria:

* serious illness requiring medical treatment
* inability to participate in physical activity due to severe disability
* history of schizophrenia, psychosis or untreated major depression
* unwilling to commute to study site once per week
* failure to provide written informed consent

Ages: 44 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Change in body weight | 0, 6, 12, 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan Raatz, PhD, MPH, RD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center; Mindy S Kurzer, PhD, MPH, RD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arikawa AY, Kaufman BC, Raatz SK, Kurzer MS. Effects of a parallel-arm randomized controlled weight loss pilot study on biological and psychosocial parameters of overweight and obese breast cancer survivors. Pilot Feasibility Stud. 2017 Jul 10;4:17. doi: 10.1186/s40814-017-0160-9. eCollection 2018. PMID 28702218